CLINICAL TRIAL: NCT00792753
Title: A Randomized, Single Blind, Consecutive Enrollment Evaluation of the Elixir Novolimus-Eluting Coronary Stent System With Durable Polymer Compared to the Medtronic Endeavor Zotarolimus-Eluting Coronary Stent System in the Treatment Of Patients With De Novo Native Coronary Artery Lesions And A Randomized, Consecutive Enrollment Evaluation of the Elixir Novolimus-Eluting Coronary Stent System With Bioabsorbable Polymer Compared to the Medtronic Endeavor Zotarolimus-Eluting Coronary Stent System in the Treatment Of Patients With De Novo Native Coronary Artery Lesions
Brief Title: Elixir Medical Clinical Evaluation of the Novolimus-Eluting Coronary Stent System: A Randomized Study "EXCELLA II STUDY"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ELX-CL-0801
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1. DESyne DES (Experimental): Test arm: Intervention with DESyne Novolimus-Eluting Coronary Stent DESyne Novolimus Stent System
  Interventions: Device: DESyne Novolimus Stent System
- 2. Medtronic Endeavor DES (Active Comparator): Control arm: Intervention with Medtronic Endeavor Zotarolimus-Eluting Coronary Stent Medtronic Endeavor Coronary Stent System
  Interventions: Device: Medtronic Endeavor Coronary Stent System
- 3. DESyne BD DES (Experimental): Test arm: Intervention with DESyne BD Novolimus-Eluting Coronary Stent DESyne BD Novolimus Stent System
  Interventions: Device: DESyne BD Novolimus Stent System

INTERVENTIONS:
Device: Medtronic Endeavor Coronary Stent System — coronary stent implantation
  Arms: 2. Medtronic Endeavor DES
Device: DESyne BD Novolimus Stent System — coronary stent implantation
  Arms: 3. DESyne BD DES
Device: DESyne Novolimus Stent System — coronary stent implantation
  Arms: 1. DESyne DES

SUMMARY:
Randomized Study To evaluate the safety and effectiveness of the Elixir Medical DESyne Novolimus-Eluting Coronary Stent System with Durable Polymer through the assessment of clinical, angiographic and IVUS endpoints as compared to the concurrently enrolled Medtronic Zotarolimus-Eluting Coronary Stent System in a randomized, single blind study of up to 200 male and female patients. In a Continued Access Registry of up to 100 patients receiving the DESyne Stent clinical-only endpoints will be evaluated.

To evaluate the safety and effectiveness of the Elixir Novolimus-Eluting Coronary Stent System with bioabsorbable polymer as compared to the Medtronic Endeavor Zotarolimus-Eluting Coronary Stent System control through clinical and angiographic endpoints.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a planned intervention of a single lesion in one or two separate major epicardial territories. Each lesion/vessel must meet the following criteria:
* De novo
* The target lesion reference site must be visually estimated to be > 2.5 mm and < 3.5 mm in diameter.
* The target vessel must be a major coronary artery or major branch with a visually estimated stenosis of > 50% and <100%.
* The visually estimated target lesion must be able to be covered by a single, 14, 18 or 28mm stent Elixir Stent or a single 14, 18, 24 or 30mm Endeavor Stent. Note that the 8mm Endeavor Stent will not be used in this study.
* Maximum lesion length is 24 mm.
* > TIMI 1 coronary flow.

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, mTOR inhibitor class drugs, cobalt chromium alloy, methacrylate or polylactide polymer, or sensitivity to contrast which cannot be adequately premedicated.
* There will be an untreated significant lesion of > 40% diameter stenosis remaining proximal or distal to the target site after the planned intervention.
* Total occlusion or TIMI 0 coronary flow in the target vessel.
* Restenosis lesion
* The proximal target vessel or target lesion is severely calcified by visual assessment.
* Aorto-ostial location, unprotected left main lesion location, or a lesion within 5 mm of the origin of the LAD or LCX.
* Lesion involvement of a significant side branch (branch diameter > 2 mm) that would be covered by stenting.
* The patient has suffered a myocardial infarction with total creatine kinase (CK) >2 times normal within the past 72 hours (exactly three days).
* The patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* The patient suffered a stroke, transient ischemic neurological attack (TIA) or significant gastrointestinal (GI) bleed within the past six months.
* The patient has renal insufficiency as determined by a creatinine of > 2.0mg/dl.
* The target lesion, or the target vessel proximal to the target lesion, contains thrombus.
* Documented left ventricular ejection fraction of < 25%.
* The patient is a recipient of a heart transplant.
* The patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion or extreme anti-coagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2008-10; Primary Completion 2011-11 (Actual); Study Completion 2014-03-08 (Actual)

PRIMARY OUTCOMES:
In-stent late lumen loss assessed by QCA | 9 months

SECONDARY OUTCOMES:
Device-oriented Composite Endpoints | 1, 6, 9, and 12 months and annually to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W Serruys, MD, PhD, Principal Investigator — Thoraxcentrum, Rotterdam, Netherlands
Locations (8):
- Monash Medical Center, Melbourne, Australia
- University Hospital Gent, Ghent, Belgium
- Instituto Dante Pazzanese, São Paulo, Brazil
- Universitäres Herz- und Gefäßzentrum, Hamburg, Germany
- Thoraxcentrum, Rotterdam, Netherlands
- Auckland City Hospital, Auckland, New Zealand
- Jagiellonian University, Krakow, Poland
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Iqbal J, Verheye S, Abizaid A, Ormiston J, de Vries T, Morrison L, Toyloy S, Fitzgerald P, Windecker S, Serruys PW. DESyne novolimus-eluting coronary stent is superior to Endeavor zotarolimus-eluting coronary stent at five-year follow-up: final results of the multicentre EXCELLA II randomised controlled trial. EuroIntervention. 2016 Dec 10;12(11):e1336-e1342. doi: 10.4244/EIJY15M10_04. PMID 26465374